CLINICAL TRIAL: NCT02004964
Title: Screening of Subjects With Type I Diabetes to Determine Eligibility for Islet Transplantation
Status: Completed | Type: Observational
Sponsor: Rodolfo Alejandro (Other)
Responsible Party: Sponsor-Investigator, Rodolfo Alejandro, Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Other Study IDs: 20053135
Record Dates: First submitted 2013-11-25; First posted 2013-12-09 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Protocol to screen potential subjects for islet transplantation

DETAILED DESCRIPTION:
Subjects with Type 1 diabetes and history of severe hypoglycemia will undergo screening similar to the screening done for islet transplantation including: history; physical; chest X rays; upper GI series if history of ulcer; abdominal and pelvic ultrasound with careful attention to liver parenchyma and gallbladder; EKG; stress echocardiography if older than 35, psychological evaluation; autonomic and sensorimotor evaluation. They will also have a tuberculosis skin test (PPD), and pre-transplant laboratory tests, including: serology (for hepatitis B and C, HTLV I and II, Herpesvirus 1 and 2, CMV, EBV, Parvovirus B19, RPR and HIV); first morning urine (albumin, protein and creatinine), GFR; urinalysis and urine culture; CBC, chemistry, PT, PTT, INR, C-peptide (basal and stimulated), HbA1c, , lipid profile, LFTs, thyroid profile, blood typing, PRA, MHC determination, auto-antibodies (GAD65, IA2 and insulin), and if male, prostate specific antigen (PSA). Severity of glucose lability and hypoglycemia unawareness is assessed with Clarke score, Lability index, Mage and hypoglycemia score.

I

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 65 years of age
2. Patients with type 1 diabetes mellitus for more than 5 years duration
3. Body Mass Index (BMI)
4. Fulfill one or more of the following:

1. Manifest signs and symptoms that are severe enough to be incapacitating. Incapacitating signs and symptoms include hypoglycemic episodes requiring assistance by others and hypoglycemia unawareness, (the inability to recognize low blood glucoses; glucoses <54 mg/dl); and/or 2. Patients with poor diabetes control (HbA1c > 8.0% but < 12%), despite intensive insulin therapy, as defined by: self monitoring of blood glucose ≥ 4 times/day, and multiple insulin injections (≥ 3/day) or insulin pump, and close monitoring of blood glucose control by an Endocrinologist.; and/or 3. Progressive diabetic complications.

Exclusion Criteria: Potential candidates will be excluded as per following criteria:

1. Age <18 or >65 years;
2. Duration of diabetes <5 years;
3. Do not have a physician that is monitoring diabetes for > 6 months;
4. Body Mass Index >30
5. Weight >80 kg;
6. Insulin requirement >1.0 u/kg/d;
7. HbA1C >12%;
8. Stimulated or basal C-peptide >0.3 ng/ml;
9. Iohexol GFR<80
10. Macroalbuminuria (>300 mg/24 hours);
11. Anemia consistently lower than the normal range.
12. Hyperlipidemia (fasting LDL cholesterol>130mg/dl and/or fasting triglycerides >200mg/dl);
13. Abnormal liver function tests (consistently >1.5 x normal range);
14. Serological evidence of HIV, HBsAg and/or HBcAb, HBsAb without history of vaccination, HTLV-1 or HCV;
15. Negative serology for Epstein Barr virus (EBV) or evidence of acute or chronic infection (IgM≥IgG);
16. Lack of updated immunizations per current CDC guidelines (including Lack of immunization against hepatitis B, pneumococcus and influenza - during season);
17. Presence of panel reactive antibodies by flow cytometry
18. Prostate specific antigen (PSA) >4 ng/ml unless malignancy ruled out;
19. Positive tuberculin test (unless proof of adequate treatment can be provided);
20. X-ray evidence of pulmonary infection or other significant pathology;
21. Gall stones and/or portal hypertension and/or hemangioma on liver ultrasound;
22. Abnormal abdominal or pelvic ultrasound (evidence of masses that are considered suspicious for malignancy or adenopathy);
23. Active peptic ulcer disease;
24. Active infections;
25. Unstable cardiovascular status (including positive stress echocardiography if >age 35)/MI in the past 6 months/LVEF<30%)
26. Untreated or unstable proliferative diabetic retinopathy;
27. Previous/concurrent organ transplantation (except failed islet cell / pancreas transplantation);
28. Malignancy or previous malignancy;
29. Any medical condition requiring chronic use of steroids;
30. Active alcohol or substance abuse; smoking in the last 6 months;
31. Sexually active females who are not: a) post-menopausal, b) surgically sterile, or c) not using an acceptable method of contraception (oral contraceptives, Norplant, Depo-Provera, and barrier devices with spermicide are acceptable; condoms used alone are not acceptable);
32. Positive pregnancy test or intent for future pregnancy, or male subject's intent to procreate;
33. Any condition or any circumstances that makes it unsafe to undergo an islet cell transplant;
34. Psychogenically unable to comply;
35. Failed psychological evaluation.
36. Persistent leukopenia (white blood cell count <3,000/uL on more than 3 occasions)
37. Acute or chronic pancreatitis.
38. Severe or unremitting diarrhea, vomiting or othe gastrointestinal disorder potentially interfering with the ability to absorb oral medications.
39. Lymphopenia - < 1,000/uL 40 Neutropenia - <1,500/uL

41. Thrombocytopenia - <100,000/uL

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with type 1 DM
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
eligibility for islet transplantation | Baseline
  This trial has the objective to determine subject eligibility for future islet transplant trials using fasting labs (including CBC, Chemistry, PRA, auto-antibodies, coagulation panel and others); a mixed meal tolerance test, psychological evaluation and a physical exam.

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Alejandro, MD, Principal Investigator — University of Miami
Locations (1):
- Diabetes Research Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided